CLINICAL TRIAL: NCT01028170
Title: Assessing the Renal Consequences and Functional Efficacy of Low Dose Hypertonic Saline Solution and Furosemide for the Treatment of Congestive Heart Failure in a Randomized, Double Blind, Prospective Study
Brief Title: Safety and Efficacy of Low Dose Hypertonic Saline Solution and High Dose Furosemide for Congestive Heart Failure
Acronym: REaCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aspirus Heart and Vascular Institute-Research and Education (Other)
Collaborators: Aspirus Wausau Hospital (Unknown)
Responsible Party: Principal Investigator, Karen Olson, Research Manager, Aspirus Heart and Vascular Institute-Research and Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REaCH-23.07.09
Record Dates: First submitted 2009-11-27; First posted 2009-12-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Congestive Heart Failure; Renal Insufficiency
Keywords: Congestive Heart Failure; Renal Insufficiency; Cardio-renal Syndrome
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardio-Renal Syndrome | interventions — Furosemide; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide with Hypertonic Saline (Experimental): Furosemide with 150 mL of 2.4% NaCl
  Interventions: Drug: furosemide and hypertonic saline solution
- Pulse Furosemide (Active Comparator): 80-160 mg furosemide (Given over 5 min IV twice a day)
  Interventions: Drug: furosemide

INTERVENTIONS:
Drug: furosemide and hypertonic saline solution — 250-500 mg furosemide (30 min IV Q 12 hours) with 150 mL of 2.4% NaCl
  Arms: Furosemide with Hypertonic Saline
Drug: furosemide — 80-160 mg furosemide (Given over 5 min IV twice a day)
  Arms: Pulse Furosemide

SUMMARY:
The purpose of this study is to compare high dose furosemide in combination with low volume hypertonic saline solution (2.4%) with intermittent pulse dose furosemide in patients with pre treatment kidney function impairment. The hypothesis is that it will provide effective diuretic response and have a beneficial effect on preservation of renal function as compared to pulse furosemide in patients with pre-treatment renal impairment (GFR < 60 mL/min).

DETAILED DESCRIPTION:
Currently, congestive heart failure (CHF) is the fastest growing heart-related diagnosis in North America, with the chance of a person experiencing it during their lifetime around 20%. In patients with CHF, acute decompensation requiring hospitalizations are common. Patients with renal insufficiency are more susceptible to worsening of renal function or overt renal failure in relation to an episode of decompensated heart failure. Thus, there is a great need for treatment to help patients with renal dysfunction that can simultaneously protect them from further renal deterioration. Preliminary evidence indicates that hypertonic saline solution (HSS) combined with high dose loop diuretics may improve the prognosis for patients with CHF. In two separate studies, this treatment was found to alleviate symptoms of CHF, and significantly reduce hospital length of stay, as well as reduce morbidity and mortality subsequent to hospital stay. So far, available studies have demonstrated that renal function is not compromised when using HSS and high dose furosemide as a treatment for CHF. Preliminary data from our institution suggests that low volume HSS combined with high dose furosemide may be beneficial for patients with renal insufficiency.

Hypothesis:

High dose furosemide in combination with low volume HSS provides effective diuretic response and has a beneficial effect on preservation of renal function while in hospital as compared to pulse furosemide in patients with pre-treatment renal impairment (GFR < 60 mL/min).

ELIGIBILITY:
Inclusion Criteria:

* Uncompensated CHF
* Framingham Criteria for HF

  * 2 Major or
  * 1 Major 2 minor

Major criteria:

* Paroxysmal nocturnal dyspnea
* Neck vein distention
* Rales
* Radiographic cardiomegaly (increasing heart size on chest radiography)
* Acute pulmonary edema
* S3 gallop
* Increased central venous pressure (>16 cm H2O at right atrium)
* Hepatojugular reflux
* Weight loss > 4.5 kg in 5 days in response to treatment

Minor criteria:

* Bilateral ankle edema
* Nocturnal cough
* Dyspnea on ordinary exertion
* Hepatomegaly
* Pleural effusion
* Decrease in vital capacity by one third from maximum recorded
* Tachycardia (heart rate>120 beats/min.)
* No Ejection Fraction Inclusion Criteria
* GFR £ 60 mL/min
* GFR (mL/min/1.73 m2) = 186 x (Scr)-1.154 x (Age)-0.203 x (0.742 if female) x (1.212 if African American) (conventional units).
* Informed consent

Exclusion Criteria:

* Patients with Acute Coronary Syndrome
* Post -op patients within 90 days of previous surgery
* Patients currently on dialysis
* Hospice patients
* Patients < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Renal function (GFR) | 30 days

SECONDARY OUTCOMES:
Diuretic response (defined as achievement of weight within 2% of previously determined dry body weight or reaching a clinically compensated state including return of functional level to prior NYHA class as determined by the primary treating physician) | one week
Length of hospital stay | 30 days
Readmission rate | 6 months
Weight loss | one week
BNP Levels | discharge, 30 days and 6 months
Hospitalization cost analysis | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Engelmeier, MD, Principal Investigator — Aspirus Heart and Vascular Institute-Research and Education; German Larrain, MD, Study Director — Aspirus Heart and Vascular Institute-Research and Education
Locations (1):
- Aspirus Wausau Hospital, Wausau, Wisconsin, United States

REFERENCES:
- [Background] MacIntyre K, Capewell S, Stewart S, Chalmers JW, Boyd J, Finlayson A, Redpath A, Pell JP, McMurray JJ. Evidence of improving prognosis in heart failure: trends in case fatality in 66 547 patients hospitalized between 1986 and 1995. Circulation. 2000 Sep 5;102(10):1126-31. doi: 10.1161/01.cir.102.10.1126. PMID 10973841
- [Background] Lapman PG, Golduber GN, Le Jemtel TH. Heart failure treatment and renal function. Am Heart J. 2004 Feb;147(2):193-4. doi: 10.1016/j.ahj.2003.10.003. No abstract available. PMID 14760310
- [Background] Paterna S, Parrinello G, Amato P, Dominguez L, Pinto A, Maniscalchi T, Cardinale A, Licata A, Amato V, Licata G, Di Pasquale P. Tolerability and efficacy of high-dose furosemide and small-volume hypertonic saline solution in refractory congestive heart failure. Adv Ther. 1999 Sep-Oct;16(5):219-28. PMID 10915397
- [Background] Licata G, Di Pasquale P, Parrinello G, Cardinale A, Scandurra A, Follone G, Argano C, Tuttolomondo A, Paterna S. Effects of high-dose furosemide and small-volume hypertonic saline solution infusion in comparison with a high dose of furosemide as bolus in refractory congestive heart failure: long-term effects. Am Heart J. 2003 Mar;145(3):459-66. doi: 10.1067/mhj.2003.166. PMID 12660669
- [Background] Paterna S, Di Pasquale P, Parrinello G, Fornaciari E, Di Gaudio F, Fasullo S, Giammanco M, Sarullo FM, Licata G. Changes in brain natriuretic peptide levels and bioelectrical impedance measurements after treatment with high-dose furosemide and hypertonic saline solution versus high-dose furosemide alone in refractory congestive heart failure: a double-blind study. J Am Coll Cardiol. 2005 Jun 21;45(12):1997-2003. doi: 10.1016/j.jacc.2005.01.059. PMID 15963399
- See also: Website for sponsoring organization — http://www.carefoundation.org